CLINICAL TRIAL: NCT06825650
Title: Investigation of the Cultural Adaptation, Validity, and Reliability of the Turkish Version of the Central Aspects of Pain (CAP) Questionnaire
Brief Title: Investigation of the Cultural Adaptation, Validity, and Reliability of the Turkish Version of the CAP Questionnaire
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Other Study IDs: SBA 24/997
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis; Back Pain; Fibromyalgia
Keywords: nociplastic pain; central sensitization; back pain; osteoarthritis; fibromyalgia; pain
MeSH Terms: conditions — Osteoarthritis; Back Pain; Fibromyalgia; Nociplastic Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Individuals with osteoarthritis
  Interventions: Other: Questionnaire study
- Individuals with back pain
  Interventions: Other: Questionnaire study
- Individuals with fibromyalgia
  Interventions: Other: Questionnaire study

INTERVENTIONS:
Other: Questionnaire study — Questionnaire application
  Other Names: CAP questionnaire

SUMMARY:
The "CAP questionnaire," developed by modifying the CAP-Knee questionnaire to assess potential nociplastic pain features in painful musculoskeletal disorders, has been described. The "CAP questionnaire" is used in people with musculoskeletal pain and diagnostic subgroups of osteoarthritis, back pain, and fibromyalgia. There is no Turkish version of the CAP questionnaire. This study aims to investigate the cultural adaptation, validity, and reliability of the Turkish version of the "CAP questionnaire."

DETAILED DESCRIPTION:
Chronic pain is a symptom shared by many musculoskeletal conditions, even when disease management is optimized. Musculoskeletal pathologies are reported to be an essential therapeutic target in pain management. However, these pathologies often do not adequately explain the pain or the reason for its persistence.

Central sensitization is the increased sensitivity of Central Nervous System (CNS) neurons to a standard nociceptive input. Pain that increases in intensity and distribution beyond that explained by musculoskeletal pathology has been termed "nociplastic pain." Measuring these CNS aspects of pain is a prerequisite for understanding their mechanistic basis and predicting future pain and responses to treatment. Chronic pain is associated with CNS dysfunction in several areas, including depression, anxiety, pain catastrophizing, cognitive dysfunction, sleep disturbance, and fatigue. Considering the increasing importance of assessing mood-related pain (nociplastic pain) The "CAP questionnaire," developed by modifying the CAP-Knee questionnaire to assess potential nociplastic pain features in painful musculoskeletal disorders, has been described.

ELIGIBILITY:
Inclusion Criteria:

* People with musculoskeletal pain and in diagnoses with OA, back pain, or FM
* Above 18 years of age
* Informed consent of the participant

Exclusion Criteria:

* Diagnosis of uncontrolled/other clinically significant diseases (chronic obstructive pulmonary disease, congestive heart failure, endocrine system diseases, neurological, psychological diseases, etc.)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who come to the university hospital for routine controls.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2027-11-28 (Estimated); Study Completion 2027-11-28 (Estimated)

PRIMARY OUTCOMES:
Central Aspects of Pain Questionnaire (CAP) | Three months
  The CAP questionnaire consists of eight items assessing each of the eight characteristics linked to the central mechanisms of knee pain over the past week. These items assess neuropathic-like pain, fatigue, cognition, catastrophizing, anxiety, depression, sleep, and widespread pain.

SECONDARY OUTCOMES:
BETY-Biopsychosocial Questionnaire | Three months
Hospital Anxiety Depression Scale (HADS) | Three months
Health Assessment Questionnaire (HAQ) | Three months
Pain Catastrophizing Scale (PCS) | Three months
Central Sensitisation Inventory (CSI) | Three months
Short-Form of McGill's Pain Questionnaire | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Will not be shared to protect the data of individuals